CLINICAL TRIAL: NCT02882971
Title: Objective Pain Score for Chronic Pain Clinic Patients
Status: Completed | Type: Observational
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Jill Eckert, Associate Professor of Anesthesiology and Pain Medicine, Milton S. Hershey Medical Center
Other Study IDs: STUDY00003685
Record Dates: First submitted 2016-03-22; First posted 2016-08-30 (Estimated); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Chronic Pain
Keywords: chronic pain; rating scale
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Pain Assessment — To create an objective observational pain scoring system and validate.

SUMMARY:
Currently, there is no observational pain scale for use in the outpatient setting for adult patients. An observational pain scale can allow for objective measurement of pain in patients over time and after treatment without the bias associated with self-report. Currently chronic pain patients are asked to rate their pain many times throughout their care, often over years. This introduces a bias in reporting as a pain a person is currently experiencing will seem more severe then a remembered pain event. A behavioral pain scale would allow for an objective measurement of pain that is reliable across multiple raters and comparable over time, which can help in judging the success of pain treatments.

DETAILED DESCRIPTION:
This is a prospective observational study. No changes in therapy will be initiated due to the information gathered by its protocol. All medical decisions will be based on the management of the clinical team. Data will be gathered during the subject's clinical visit, from the subject, and from the nursing staff caring for the subject.

The Chronic Pain Behavioral Pain Scale for Adults was developed by the research team based on behavior pain scales used in other populations and the clinical expertise of Chronic Pain specialists in the Hershey Medical Center Chronic Pain department.

Patients will be scored on the Chronic Pain Behavioral Pain Scale for Adults and the standard 11 point numeric rating scale (Jensen, Turner et al., 1996), on intake. Scoring will be done by the patient's assigned nurse and a member of the research team, at the time when the numeric pain score is typically obtained. The patient will be scored again on both the Chronic Pain Behavioral Pain Scale for Adults and the standard numeric rating pain scale at the conclusion of their procedure, again at the time when the numerical pain score is typically obtained. Scoring will again be done by the patient's assigned nurse and a member of the research team. The Chronic Pain Behavioral Pain Scale for Adults will be tested for inter-rater reliability using the paired scores from the nurse and researcher for each subject. Concurrent Validity will be measured using comparison between the numeric rating scale and the behavioral pain scale on each subject at each time point. Construct validity will be measured by comparing the behavioral pain score before and after the interventional pain treatment.

For training purposes, the assigned nurse and research team member will be provided a copy of the "Chronic Pain Behavioral Pain Scale for Adults" chart to be utilized during their patient encounters. Each team member will be individually instructed in the use of the scale immediately preceding their first use of the scales. This training will include a discussion of the elements, the definition of behaviors, and the use of the scoring system.

ELIGIBILITY:
Inclusion Criteria:

1. Adults age 18-75
2. Patients able to self-report their pain using a validated pain scale
3. Patients of the chronic pain clinic who will be receiving a pain treatment procedure
4. English speaking
5. Received and signed a consent to participate in the study

Exclusion Criteria:

1. Pregnant and lactating women
2. Patient with chronic malignant pain
3. Patients less than 18
4. Patient older than 75
5. Patients with dementia
6. Non-English speaking patients
7. Patients unable to do a self-report pain scale
8. Uncontrolled psychiatric conditions
9. Uncontrolled substance abuse issues
10. Patient's lost to follow-up
11. Patients who don't wish to participate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults between the ages of 18-75 that are able to self-report their pain level using a validated pain scale.
Sampling Method: Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Patient's pre-procedure pain score using the Chronic Pain Behavioral Scale for Adults. | Within 30 minutes prior to intervention designed to alleviate pain
  2 observers will use the new Chronic Pain Behavioral Scale for Adults to measure the patient's pain before a procedure to alleviate pain.
Patient's pre-procedure pain score using the standard 11-point numerical rating scale. | Within 30 minutes prior to an intervention designed to alleviate pain
  The patient will be asked to rate their pain, using the standard 11-point numerical rating scale, before a procedure to alleviate pain.

SECONDARY OUTCOMES:
Patient's post-procedure pain score using the Chronic Pain Behavioral Scale for Adults. | Within 3 h after an intervention designed to alleviate pain
  2 observers will use the new Chronic Pain Behavioral Scale for Adults to measure the patient's pain before a procedure to alleviate pain.
Patient's post-procedure pain score using the standard 11-point numerical rating scale. | Within 3 h after an intervention designed to alleviate pain
  The patient will be asked to rate their pain, using the standard 11-point numerical rating scale, before a procedure to alleviate pain.

CONTACTS AND LOCATIONS:
Overall Officials: Jill Eckert, DO, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jensen MP, Turner LR, Turner JA, Romano JM. The use of multiple-item scales for pain intensity measurement in chronic pain patients. Pain. 1996 Sep;67(1):35-40. doi: 10.1016/0304-3959(96)03078-3. PMID 8895229
- [Derived] Pace AK, Bruceta M, Donovan J, Vaida SJ, Eckert JM. An Objective Pain Score for Chronic Pain Clinic Patients. Pain Res Manag. 2021 Feb 8;2021:6695741. doi: 10.1155/2021/6695741. eCollection 2021. PMID 33628355